CLINICAL TRIAL: NCT01714960
Title: Safety and Tolerability of MRZ-99030 Eye Drops in Healthy Volunteers and Glaucoma Patients
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Merz Pharmaceuticals GmbH (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MRZ99030_1001_1; 2012-002664-26 (EudraCT Number)
Record Dates: First submitted 2012-10-24; First posted 2012-10-26 (Estimated); Last update posted 2014-01-29 (Estimated); Status verified 2014-01

CONDITIONS: Healthy Volunteers and Glaucoma Patients

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Healthy volunteers low dose (Experimental): MRZ-99030 eye drops (5mg/mL), 1-3 drops three times per day, duration: 16 days.
  Interventions: Drug: MRZ-99030 eye drops 5mg/mL
- Healthy volunteers high dose (Experimental): MRZ-99030 eye drops (20mg/mL), 1-3 drops three times per day, duration: 16 days.
  Interventions: Drug: MRZ-99030 eye drops 20mg/mL
- Glaucoma patients (Experimental): MRZ-99030 eye drops (20mg/mL), 1-3 drops three times per day, duration: 16 days.
  Interventions: Drug: MRZ-99030 eye drops 20mg/mL
- Placebo (Placebo Comparator): Placebo eye drops, 1-3 drops three times per day, duration: 16 days.
  Interventions: Drug: Placebo to MRZ-99030 eye drops

INTERVENTIONS:
Drug: MRZ-99030 eye drops 5mg/mL
  Arms: Healthy volunteers low dose
Drug: MRZ-99030 eye drops 20mg/mL
  Arms: Glaucoma patients; Healthy volunteers high dose
Drug: Placebo to MRZ-99030 eye drops
  Arms: Placebo

SUMMARY:
* To assess the safety and tolerability of repeat dose topical administration of MRZ-99030 Ophthalmic Solution with ascending doses in healthy subjects (stage 1) and glaucoma subjects (stage 2).
* To assess plasma pharmacokinetics and urine concentration of MRZ- 99030 and its metabolite MRZ-9499 after single and repeat dose topical administration of MRZ-99030 Ophthalmic Solution.

ELIGIBILITY:
Inclusion Criteria:

For stage 1:

- Healthy volunteers

For stage 2:

- Glaucoma patients

Exclusion Criteria:

For stage 2:

- Any relevant eye disease other than glaucoma

Ages: 35 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2012-10; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Incidence of adverse events | Day 1 up to day 23

SECONDARY OUTCOMES:
Area under the curve (AUC) | Day 1 to day 17
Maximal plasma concentration (Cmax) | Day 1 to day 17

CONTACTS AND LOCATIONS:
Overall Officials: Medical Expert, Study Director — Merz Pharmaceuticals GmbH
Locations (1):
- Parexel International GmbH, Early Phase Clinical Unit, Berlin, Germany